CLINICAL TRIAL: NCT01938144
Title: Three-day Clinical Evaluation Of The Efficacy And Safety Of Two Ibuprofen Combination Products For The Symptomatic Treatment Of The Common Cold And Flu: A Multicenter Study
Brief Title: Evaluation of the Efficacy and Safety of Two Ibuprofen Combination Products for the Treatment of the Common Cold and Flu in Latin America
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B3971002; U1111-1147-8736 (Other: Alias Study Number)
Record Dates: First submitted 2013-09-04; First posted 2013-09-10 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Common Cold
Keywords: Common cold; efficacy; symptoms; Wisconsin Upper Respiratory Symptom Survey - 21; ibuprofen; phenylephrine; pseudoephedrine
MeSH Terms: conditions — Common Cold | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment A (Experimental): IBU 200 mg/ PE 10 mg
  Interventions: Drug: Advil Congestion Relief
- Treatment B (Experimental): IBU 200 mg/ PE 10 mg/CHLOR 4 mg
  Interventions: Drug: Advil Allergy and Congestion Relief
- Treatment C (Active Comparator): Acetaminophen 500 mg
  Interventions: Drug: Paracetamol

INTERVENTIONS:
Drug: Advil Congestion Relief — Orally adminstered, 200 mg Ibuprofen/10 mg Phenylephrine tablet, 4x/day, up to 8 doses.
  Arms: Treatment A
Drug: Advil Allergy and Congestion Relief — Orally adminstered, 200 mg Ibuprofen/10 mg Phenylephrine/4 mg Chlorpheniramine tablet, 4x/day, up to 8 doses.
  Arms: Treatment B
Drug: Paracetamol — Acetaminophen 500 mg, 4x/day, up to 8 doses.
  Arms: Treatment C

SUMMARY:
This is a multicenter, prospective, randomized, double-blind, triple-dummy, parallel group, comparative, study designed to evaluate the efficacy of Ibuprofen (IBU) 200 mg/ Phenylephrine (PE) 10 mg and IBU 200 mg/ PE 10 mg/ Chlorpheniramine (CHLOR) 4 mg on the relief of symptoms of the common cold and flu. The reference product that the active treatments will be compared to is paracetamol (PARA) 500 mg.

ELIGIBILITY:
Inclusion Criteria:

Male and female subjects who are 18 years old or older at the time of screening.

Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Subjects must present with a score of 5 of higher for at least 2 of the following 6 symptoms: runny nose, plugged nose, sneezing, sore throat, scratchy throat, or head congestion on the WURSS-21 assessment, within 36 hours of onset of symptoms.

Exclusion Criteria:

Anyone with a history of chronic allergic rhinitis or asthma at the time of the screening visit, or with history of chronic recurrent airway disease, infections, or frequent complications of colds (otitis media, sinusitis, or bronchitis)

Subjects taking any prescription or non-prescription drug, within the last 7 days prior to the screening, with which the administration of IBU, PE, CHLOR, or APAP is contraindicated, may increase the risk associated with study participation, or may interfere with the interpretation of study results, in the judgment of the Investigator.

Subjects currently taking a monoamine oxidase (MAO) inhibitor, or has taken an MAO inhibitor within 2 months of screening.

Subjects currently taking a serotonin-selective reuptake inhibitor (SSRI), tricyclic antidepressant (TCA), barbiturate, or any other neuroleptic, or has taken an SSRI, TCA, barbiturate, or any other neuroleptic within 14 days of screening.

Subjects with a hypersensitivity to IBU, PE, or CHLOR or APAP.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-04; Primary Completion 2016-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the sum of 6 of the most common cold and flu symptoms (runny nose, plugged nose, sneezing, sore throat, scratchy throat, and head congestion), averaged over the treatment period assessed using the Wisconsin Upper Respiratory | 2 Days
  The severity of cold/flu symptoms will be determined by the subject's response to the Wisconsin Upper Respiratory Symptom Survey, which includes questions related to the signs and symptoms of cold and flu, as well as Quality of Life Measures.
Symptom Survey - 21 | 2 Days
  The severity of cold/flu symptoms will be determined by the subject's response to the Wisconsin Upper Respiratory Symptom Survey, which includes questions related to the signs and symptoms of cold and flu, as well as Quality of Life Measures.

SECONDARY OUTCOMES:
Change from baseline in the sum of all 10 common cold and flu symptoms, averaged over the treatment period. | 2 Days
  The severity of cold/flu symptoms will be determined by the subject's response to the Wisconsin Upper Respiratory Symptom Survey, which includes questions related to the signs and symptoms of cold and flu, as well as Quality of Life Measures.
Change from baseline in the sum of 6 of the most common symptoms at each assessment (PM day 1, AM and PM day 2) | 2 Days
  The severity of cold/flu symptoms will be determined by the subject's response to the Wisconsin Upper Respiratory Symptom Survey, which includes questions related to the signs and symptoms of cold and flu, as well as Quality of Life Measures.
Symptom relief since taking the first dose | 1 hours
  One Hour Assessment of Relief question following the first dose

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B3971002&StudyName=Evaluation%20of%20the%20Efficacy%20and%20Safety%20of%20Two%20Ibuprofen%20Combination%20Products%20for%20the%20Treatment%20of%20the%20Common%20Cold%20and%20Flu%20in%20Latin%20